CLINICAL TRIAL: NCT02935166
Title: INNOTORIO: Innovations in the Training of the Inspiratory Muscles on Patients With Chronic Obstructive Pulmonary Disease: Design of a Digital Dual Valve and Evaluation of a New High-intensity Training Scheme of Short Duration.
Brief Title: Innovations in Respiratory Muscles Training in Patients With Chronic Obstructive Pulmonary Disease. (INNOTORIO)
Acronym: INNOTORIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 656656933786
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: COPD; Respiratory Muscles; Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Uncharged (Placebo Comparator): Respiratory muscle training: placebo General High Intensity Training (30 minutes in cycle ergometer) and placebo respiratory muscle training: This training group performed with the valve Orygen® uncharged (placebo effect). Performing 10 consecutive inspirations (5 series) two times a day during 3 weeks.
  Interventions: Other: Respiratory muscle training
- Inspiratory (Active Comparator): Respiratory muscle training: Inspiratory General Training (30 minutes in cycle ergometer) and high intensity inspiratory muscle training: The inspiratory training was conducted with the Orygen® valve. Inspiratory training load was defined as maximum and patient tolerance that would perform 10 consecutive inspirations (5 series) two times a day, during 3 weeks.
  Interventions: Other: Respiratory muscle training
- Inspiratory and expiratory (Active Comparator): Respiratory muscle training: Inspiratory and expiratory General High Intensity Training (30 minutes in cycle ergometer) and inspiratory and expiratory training: The inspiratory and expiratory training was conducted with the Orygen® valve. Loading inspiratory and expiratory training was defined as maximum and patient tolerance. This was the optimal load that would allow the patient to perform 10 consecutive inspirations (5 sessions) 2 times a day,during 3 weeks.
  Interventions: Other: Respiratory muscle training

INTERVENTIONS:
Other: Respiratory muscle training — General high-intensity training consists in maximum effort intervals of 30 seconds duration against an equivalent resistance 0.075 kg / kg of body mass followed by a recovery period of 4 minutes cycle ergometer; the total duration was 3 weeks. They were made in this regard, five weekly sessions of 30 minutes per session, Additionally, randomly, the patients were divided into one of 3 possible groups of respiratory training, which consisted of 5 sets of 10 full breaths (inspiration and expiration) in the morning and afternoon during 3 weeks.

SUMMARY:
Respiratory muscle weakness and fatigue are related to clinical deterioration in patients with Chronic Obstructive Pulmonary Disease (COPD). Respiratory muscle training (RMT) is a key therapeutic strategy in these patients. It is necessary therefore to increase its dissemination on a large scale, improve patient´s adherence and optimize the control of the implementation of training. The aim of this project was to design a RMT device including light and sound incentives, digital registration application and analysis of the training sessions, and studying the effectiveness of a new shortened RMT scheme of high intensity that could provide added value to enhance the implementation of training in patients with COPD. From an operational point of view, researches were organized into three packages of complementary work focused on the design of a new portable dual valve with electronic lighting and auditory incentives components. The conceptualization and design of a software to analyze the performance and individual continuous use of the valve, and the evaluation of the feasibility, safety and efficacy of a shortened schedule of respiratory muscle training in adult patients with COPD were realized.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis from moderate to severe COPD muscle weakness inspiratory Must be able to do exercises

Exclusion Criteria:

* Positive bronchodilator response Cardiovascular, neuromuscular, or metabolic disease Hospital admission for any pathology in the last two months have completed a rehabilitation program in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Respiratory muscle strength assessed by Maximun Respiratory Pressure | From baseline to 3 weeks
  Defined as the ability to make a maximum respiratory effort, it was assessed using the MicroRPM® device. This test is to generate the maximum inspiratory pressure (from residual volume) and expiratory (from total lung capacity) against a road or occluded team, performing the maneuver by keeping the mouth and nose occluded.
Change in Exercise Capacity assessed by cardiopulmonary exercise testing | From baseline to 3 weeks
Change in Quality of life assessed by Quality of life Short Form 36 questionnaire | From baseline to 3 weeks

SECONDARY OUTCOMES:
Change in Exercise Capacity assessed by Six minutes walking Test | From baseline to 3 weeks
Change in Respiratory function assessed by spirometry | From baseline to 3 weeks

IPD SHARING:
Plan to Share IPD: Yes